CLINICAL TRIAL: NCT02750163
Title: Circulating Free Hemoglobin and Microcirculation After Administration of Paracetamol in Febrile Septic Patient
Status: Completed | Type: Observational
Sponsor: Università Politecnica delle Marche (Other)
Responsible Party: Principal Investigator, Abele Donati, MD, Associate Professor, Università Politecnica delle Marche
Other Study IDs: FreeHb
Record Dates: First submitted 2016-04-16; First posted 2016-04-25 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-04

CONDITIONS: Sepsis and Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Acetaminophen

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Dosage of free hemoglobin; dosage of oxidative markers as F2-isoprostane F2 and-isoflurane, sindecan-1, heparasulfate and hyaluronic acid, endothelin-1, plasma assay of NO, reduced glutathione, haptoglobin and hemopexin, PD-1/PD-L1.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: paracetamol — Paracetamol will be given to febrile septic patients

SUMMARY:
The aim of this study is to evaluate the effect of Acetaminophen on the main parameters of microcirculation, on the plasmatic levels of free hemoglobin/oxidative stress markers and on the expression of PD1/Pd-L1, in pyrexial septic patient.

DETAILED DESCRIPTION:
It has been established that plasma levels of extra-cellular free hemoglobin increased significantly in patients with certain disease, including sickle cellular disease, or undergoing invasive treatments, like coronary bypass surgery, blood transfusions and hemodialysis.

In all these conditions, high levels of free hemoglobin were associated with poor outcome and with serious complications such as acute renal failure and myocardial infarction.

In the animal model of sepsis, increased values of plasma free hemoglobin has been related to increased mortality, especially if a concomitant lack of haptoglobin and hemopexin coexists.

It is likely that the release of free hemoglobin in the blood of septic patient is attributable to changes in the membrane of red blood cells.

These changes have been recognized in humans as a source of damage of the vascular endothelium and consumption of free radical scavenger systems.

It has been hypothesized that the extracellular hemoglobin, when the protective mechanism have been saturated, causes - trough reaction with NO - the formation of nitrate and lipids peroxidation and boosts the immune response mediated by the monocyte -macrophage system.

It is also liable for a condition of endothelial dysfunction and NO resistance that could impair the microcirculation.

Our previous work showed that higher levels of free hemoglobin resulted in a significant reduction in the density of the microcirculation in septic patients undergoing blood transfusions.

On animal model Paracetamol (or acetaminophen), drug commonly used for its analgesic and antipyretic effects, demonstrated strong efficacy in preventing oxidative damage and protection of renal damage in the context of increased levels of plasma free hemoglobin (as in Rhabdomyolysis and myoglobulinemie).

This effect is attributed to the ability of the Paracetamol to cross react with either nitric oxide synthase (NOS) by increasing the synthesis of NO, and with cyclooxygenase (COX), by inhibiting the synthesis of prostaglandin I2 (PGI2-antiplatelet and vasodilator effect) without interfering with the production of Thromboxane A2 (TXA2-powerful vasoconstrictor and pro-thrombogenic) causing an imbalance of endovascular homeostasis.

The increased oxidative stress produced by sepsis is also responsible of glycocalix damage, the thin layer that lines the surface of endothelium in contact with the blood and increased the free hemoglobin.

ROS are also responsible to up-regulation of Programmed Death-1 related molecules (PD-1/PD-L1) that render T cells susceptible to inhibitory modulation, inability to proliferate and reduced capacity to clear bacteria, inducing "immunosuppression" and more difficult recovery from septic shock. PD-1/PD-L1 system has been recently studied as potential predictor of mortality and active player in resolution of sepsis-induced Acute Lung Injury.

Finally, a recent study on septic patient showed an increased mortality in people with elevated values of free hemoglobin versus patients without this increase, and the efficacy of of Paracetamol to reduce the concentration of F2- isoprostane (marker of oxidative stress), associated with lower risk of death.

This effect was lost in the cohort of septic patients without free hemoglobin registered.

Aim of this study is to evaluate the effect of paracetamol administration on the microcirculation, on the plasmatic levels of free hemoglobin/oxidative stress markers and on the expression of PD1/Pd-L1, in pyrexial septic patient. Paracetamol is given only on the basis of a clinical indication, not because of the study and in our institution paracetamol is the drug of choice to treat fever.

When there are inclusion criteria (febrile septic patient) and no exclusion criteria, and patient is going to receive paracetamol, informed consent will be taken. When the neurological conditions do not permit, relatives will be informed and the patients will still included in the protocol. The informed consent will be taken when the patient clinical condition permits it.

Before the administration of the drug, at the end of infusion and after 30 minutes after infusion, the main parameters of the sublingual microcirculation will be monitored, using the the incident dark field imaging technique (IDF), including an assessment of glycocalyx, Near InfraRed (NIRS) parameters with the vascular occlusion test (VOT), vital signs and the dosage of any infusion of vasoactive drug.

Demographic and clinical records will be collected at T0 and T1. Acute lung injury will be investigated through gas analytical and laboratory data at the same timepoints.

Arterial blood samples will be collected at T0 and 2 hours after the infusion of Acetaminophen (that will represent T2). Blood will be immediately centrifuged and plasma and serum samples will be stored at -70°C for subsequent analysis. We will measure: fHb levels, markers of oxidative damage (F2-isoprastane and F2-isoflurane), of endothelial cell injury (endothelin-1) and glycocalyx damage (sindecan-1, heparasulfate), PD-1/PD-L1.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sepsis, severe sepsis and septic shock with high body temperature that need administration of Paracetamol and which have previously monitored blood pressure and have a central venous catheter in place.

Exclusion Criteria:

* age < 18 years
* pregnancy
* hemodialysis
* hemolysis of the blood sample
* use of Paracetamol in the previous 12 hours
* conditions that do not allow the possibility of getting a monitoring of sublingual microcirculation (maxillofacial trauma, serious inability to jaw, copious blood loss or secretions from the mouth)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 patients with sepsis or septic shock
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-06-05 (Actual)

PRIMARY OUTCOMES:
Perfused Vessel Density (PVD) | 30 minutes
  The perfused vessel density (PVD), unit of measure mm/mm2, is detected in vivo by Incident Dark Field Imaging at sublingual microcirculation. It represents the quantity of well perfused vessels at microcirculatory level.

SECONDARY OUTCOMES:
StO2 upload | 30 minutes
  StO2 upslope (%/min) is measured with Near InfraRed Spectroscopy at the tenar muscle. It represents the velocity of the recovery of the tissue oxygen saturation after a short period of ischemia of the hand, the Vascular Occlusion Test.
Microcirculatory flow index (MFI) | 30 minutes
  Microcirculatory Flow Index detected in vivo by Incident Dark Field Imaging at sublingual microcirculation. It represents the quality of blood flow at microcirculatory level.

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Ospedali Riuniti Ancona - Università Politecnica delle Marche, Ancona, Italy

REFERENCES:
- [Derived] Scorcella C, Domizi R, Amoroso S, Carsetti A, Casarotta E, Castaldo P, D'angelo C, Damiani E, Gasparri F, Donati A, Adrario E. Pharmacogenetics in critical care: association between CYP3A5 rs776746 A/G genotype and acetaminophen response in sepsis and septic shock. BMC Anesthesiol. 2023 Feb 16;23(1):55. doi: 10.1186/s12871-023-02018-y. PMID 36797680